CLINICAL TRIAL: NCT07352553
Title: Non-invasive Brain Stimulation for Postherpetic Neuralgia: A Prospective, Randomized, Sham-Controlled Study
Brief Title: Brain Stimulation for Postherpetic Neuralgia: A Randomized Sham-Controlled Trial
Acronym: PHN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang，MD, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-IRB202512160
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Stimulation + Usual Care (Experimental): Participants receive brain stimulation in addition to usual pharmacological care for postherpetic neuralgia. Brain stimulation is delivered once daily for 30 minutes for 10 consecutive days.
  Interventions: Device: Non-invasive transcranial stimulation
- Sham Stimulation + Usual Care (Sham Comparator): Participants receive sham stimulation in addition to usual pharmacological care. Electrodes are applied once daily for 30 minutes for 10 consecutive days; after an initial brief stimulation to mimic sensation, the output is turned off.
  Interventions: Device: Sham Non-invasive transcranial stimulation

INTERVENTIONS:
Device: Non-invasive transcranial stimulation — Non-invasive transcranial stimulation is delivered once daily for 30 minutes for 10 consecutive days. Stimulation is administered using a multi-channel battery-powered device with five circular Ag/AgCl electrodes; current output is monitored in real time for safety.
  Arms: Brain Stimulation + Usual Care
Device: Sham Non-invasive transcranial stimulation — Sham procedure with identical electrode placement and session duration (30 minutes once daily for 10 consecutive days). After an initial brief stimulation to mimic sensation, the current output is turned off.
  Arms: Sham Stimulation + Usual Care

SUMMARY:
Pharmacotherapy is the cornerstone of Postherpetic Neuralgia (PHN) management. First-line treatments for PHN include antiviral agents (e.g., acyclovir, valacyclovir, famciclovir, and brivudine), centrally acting antiepileptic drugs (pregabalin and gabapentin), antidepressants (duloxetine and venlafaxine), and peripherally acting sodium-channel blockers (lidocaine patches).

In recent years, substantial progress has been made in the prevention and treatment of PHN, including early and active antiviral therapy (acyclovir, valacyclovir, famciclovir, brivudine, etc.), analgesic therapy (calcium-channel modulators such as pregabalin and gabapentin; tricyclic antidepressants such as amitriptyline; and opioid analgesics), interventional procedures (e.g., radiofrequency modulation and spinal cord stimulation), and vaccination. Nevertheless, clinical outcomes remain unsatisfactory, with the incidence of refractory PHN still exceeding 50%. Adverse effects associated with certain first- and second-line medications (such as antidepressants and anticonvulsants), as well as the potential risk of opioid dependence, markedly reduce treatment adherence. This situation has compelled clinicians to continually seek new and effective therapeutic approaches for PHN.

Non-invasive transcranial stimulation, as an emerging noninvasive neuromodulation technique, enables targeted modulation of deep brain structures. Animal studies have demonstrated that it can noninvasively regulate neuronal firing in deep regions and induce long-term plasticity, while offering relatively high spatial selectivity and tissue penetration. These features suggest broad clinical potential in chronic pain and affective disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of postherpetic neuralgia (PHN) with disease duration ≥ 3 months.
* NRS pain score ≥ 4.
* Willing to receive the intervention and able to provide written informed consent.

Exclusion Criteria:

* Contraindications to electrical stimulation (e.g., intracranial metal implants, cardiac pacemaker).
* History of epilepsy, severe psychiatric disorder, or cognitive impairment.
* Pregnant or breastfeeding women.
* Unable to comply with the intervention procedures and follow-up assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity (NRS) | Baseline, Day 10 (end of treatment), 1 month, and 3 months
  Numeric Rating Scale (NRS, 0-10); change from baseline in pain intensity.

SECONDARY OUTCOMES:
Neuropathic pain symptoms | Baseline, Day 10, 1 month, 3 months
  Neuropathic Pain Symptom Inventory (NPSI); change from baseline.
Pain interference | Baseline, Day 10, 1 month, 3 months
  Brief Pain Inventory (BPI) interference subscale; change from baseline.
Health-related quality of life | Baseline, Day 10, 1 month, 3 months
  EuroQol-5 Dimension (EQ-5D); change from baseline.
Sleep quality | Baseline, Day 10, 1 month, 3 months
  Medical Outcomes Study Sleep Scale (MOS-SS); change from baseline.
Emotional status | Baseline, Day 10, 1 month, 3 months
  Generalized Anxiety Disorder-7 (GAD-7); change from baseline.Edinburgh Postnatal Depression Scale-10 (EPDS-10) or prespecified depression scale; change from baseline.Pain Catastrophizing Scale (PCS); change from baseline.
Global impression | Day 10, 1 month, 3 months
  Patient Global Impression of Change (PGIC) and Clinician Global Impression of Change (CGIC) at follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jia T, Xia J, Zhang C, Sun B, Yuan K, Liu T, Xu X, Liu J. Comparing analgesic effects of temporal interference stimulation on ventral posterolateral thalamus and high-definition transcranial alternating current stimulation on sensorimotor cortex during sustained experimental pain. Brain Stimul. 2025 May-Jun;18(3):701-703. doi: 10.1016/j.brs.2025.03.013. Epub 2025 Mar 19. No abstract available. PMID 40112912
- [Background] Grossman N, Okun MS, Boyden ES. Translating Temporal Interference Brain Stimulation to Treat Neurological and Psychiatric Conditions. JAMA Neurol. 2018 Nov 1;75(11):1307-1308. doi: 10.1001/jamaneurol.2018.2760. No abstract available. PMID 30264149
- [Background] Kurklinsky S, Palmer SC, Arroliga MJ, Ghazi SM. Neuromodulation in Postherpetic Neuralgia: Case Reports and Review of the Literature. Pain Med. 2018 Jun 1;19(6):1237-1244. doi: 10.1093/pm/pnx175. PMID 29016994
- [Background] Plow EB, Pascual-Leone A, Machado A. Brain stimulation in the treatment of chronic neuropathic and non-cancerous pain. J Pain. 2012 May;13(5):411-24. doi: 10.1016/j.jpain.2012.02.001. Epub 2012 Apr 7. PMID 22484179
- [Background] Kumar K, Taylor RS, Jacques L, Eldabe S, Meglio M, Molet J, Thomson S, O'Callaghan J, Eisenberg E, Milbouw G, Buchser E, Fortini G, Richardson J, North RB. The effects of spinal cord stimulation in neuropathic pain are sustained: a 24-month follow-up of the prospective randomized controlled multicenter trial of the effectiveness of spinal cord stimulation. Neurosurgery. 2008 Oct;63(4):762-70; discussion 770. doi: 10.1227/01.NEU.0000325731.46702.D9. PMID 18981888
- [Background] Sears NC, Machado AG, Nagel SJ, Deogaonkar M, Stanton-Hicks M, Rezai AR, Henderson JM. Long-term outcomes of spinal cord stimulation with paddle leads in the treatment of complex regional pain syndrome and failed back surgery syndrome. Neuromodulation. 2011 Jul-Aug;14(4):312-8; discussion 318. doi: 10.1111/j.1525-1403.2011.00372.x. Epub 2011 Jul 7. PMID 21992424
- [Background] Shrestha M, Chen A. Modalities in managing postherpetic neuralgia. Korean J Pain. 2018 Oct;31(4):235-243. doi: 10.3344/kjp.2018.31.4.235. Epub 2018 Oct 1. PMID 30310548
- [Background] van Hecke O, Austin SK, Khan RA, Smith BH, Torrance N. Neuropathic pain in the general population: a systematic review of epidemiological studies. Pain. 2014 Apr;155(4):654-662. doi: 10.1016/j.pain.2013.11.013. Epub 2013 Nov 26. PMID 24291734
- [Background] Holmes D. The pain drain. Nature. 2016 Jul 14;535(7611):S2-3. doi: 10.1038/535S2a. No abstract available. PMID 27410529
- [Background] Scholz J, Finnerup NB, Attal N, Aziz Q, Baron R, Bennett MI, Benoliel R, Cohen M, Cruccu G, Davis KD, Evers S, First M, Giamberardino MA, Hansson P, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Nurmikko T, Perrot S, Raja SN, Rice ASC, Rowbotham MC, Schug S, Simpson DM, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ, Barke A, Rief W, Treede RD; Classification Committee of the Neuropathic Pain Special Interest Group (NeuPSIG). The IASP classification of chronic pain for ICD-11: chronic neuropathic pain. Pain. 2019 Jan;160(1):53-59. doi: 10.1097/j.pain.0000000000001365. PMID 30586071